CLINICAL TRIAL: NCT05222880
Title: Evaluation of a Daily Disposable Silicone Hydrogel Multifocal Contact Lens in Myopes and Hyperopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6477
Record Dates: First submitted 2022-01-04; First posted 2022-02-03 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TEST Lens (Experimental): Eligible subjects who are habitual soft contact lens wearers will be given the TEST Lens for the duration of the study.
  Interventions: Device: JJVC Investigational Multifocal Contact Lenses manufactured in senofilcon A C3

INTERVENTIONS:
Device: JJVC Investigational Multifocal Contact Lenses manufactured in senofilcon A C3 — TEST Lens

SUMMARY:
This is a single-masked, single-arm, dispensing clinical trial that will evaluate vision, eye health and fit acceptance.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be at least 40 years of age and not greater than 70 years of age at the time of consent.
4. Own a wearable pair of spectacles if required for their distance vision.
5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
6. Either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
7. The subject's distance spherical equivalent refraction (vertex corrected if ≥-4.25 D) must be in the range of -1.25 D to -5.75 D or +0.75 D to +3.25 D in each eye.
8. The subject's refractive cylinder must be ≤0.75 D in each eye.
9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens- Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
4. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, peripheral iridotomy/iridectomy, cataract surgery, retinal surgery, etc.).
5. Have a history of amblyopia, strabismus or binocular vision abnormality.
6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See section 9.1 for further examples.
7. Use of any ocular medication, with the exception of rewetting drops.
8. Have a history of herpetic keratitis.
9. Have a history of irregular cornea.
10. Have a history of pathological dry eye.
11. Have Participated in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
12. Be and employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
13. Have any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.
14. Have clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
15. Have any current ocular infection or inflammation.
16. Have any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (12):
- United States (12):
  - Vue Optical Boutique, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield Hills, Michigan
  - Eye Associates of New York, Manhattan, New York
  - Sacco Eye Group, Vestal, New York
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island
  - Optometry Group, LLC, Memphis, Tennessee
  - Vision Optique, Houston, Texas
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 140 subjects were enrolled in this study. Of those enrolled, 139 subjects were dispensed at least one study lens, while 1 subject failed to meet all eligibility criteria. Of those dispensed, 136 subjects completed the study while 3 subjects were discontinued.
Groups:
- Test (Senofilcon A C3): Subjects randomized to receive the Test lens during the study
Period: Overall Study
Arm/Group | Test (Senofilcon A C3)
Started | 139
Completed | 136
Not Completed | 3
Not completed — Unsatisfactory Visual Response due to Test Article | 1
Not completed — Withdrew Consent during Study | 1
Not completed — COVID-19 Related | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Hyperopes: Subjects were classified as Hyperopic if the distance spherical equivalent refraction was in the range of +0.75 D to +3.25 D.
- Myopes: Subjects were classified as Myopic if the distance spherical equivalent refraction was in the range of -5.75 D to -1.25 D.
- Total: Total of all reporting groups
Arm/Group | Hyperopes | Myopes | Total
Number analyzed (Participants) | 50 | 89 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (7.20) | 50.4 (6.14) | 51.7 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 66 | 111
  Male | 5 | 23 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 3 | 5
  Black or African American | 2 | 9 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  White | 44 | 75 | 119
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 89 | 139

OUTCOME MEASURES:

1. Primary Outcome: Binocular logMAR Visual Acuity
Description: Binocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance high contrast condition. At distance (4 meters), VA is assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts; while near (40 cm) and intermediate (64 cm) assessments were made using reduced Guillon-Poling charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Test (Senofilcon A C3): Subjects that wore the Test lens during the study.
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 136
LogMAR
  Distance(4m) | -0.098 (0.0854)
  Intermediate (64cm) | -0.043 (0.0797)
  Near (40cm) | 0.0797 (0.1077)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% Individually) with at least 99% statistical power, that 17 subjects were required to test the primary hypothesis for Distance; Test type: Superiority — A superiority Margin of 0.00 logMAR was used for distance; Mean Population Estimate = -0.10, 99% CI 2-sided [-0.12 to -0.08], Standard Error of Mean 0.007
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% Individually) with at least 99% statistical power, that 11 subjects were required to test the primary hypothesis for Intermediate; Test type: Superiority — A superiority Margin of 0.17 logMAR was used for Intermediate; Mean Population Estimate = -0.04, 99% CI 2-sided [-0.06 to -0.02], Standard Error of Mean 0.007
Statistical Analysis 3: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% Individually) with at least 99% statistical power, that 48 subjects were required to test the primary hypothesis for Near; Test type: Superiority — A superiority Margin of 0.17 logMAR was used for near; Mean Population Estimate = 0.07, 99% CI 2-sided [0.05 to 0.09], Standard Error of Mean 0.009

2. Primary Outcome: CLUE Vision Score
Description: Subjective vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each sphere stratum (Hyperope and Myope) was reported.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 136
Units on a scale
  Hyperopes: number analyzed (Participants) | 49
  Hyperopes | 52.30 (19.121)
  Myopes: number analyzed (Participants) | 87
  Myopes | 63.27 (19.031)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% individually) with at least 99% statistical power, that 14 subjects were required to test for superiority for CLUE vision scores for Hyperopes; Test type: Superiority — A superiority Margin of 36 CLUE Points was used for Hyperopes; Mean Population Estimate = 52.3, 99% CI 2-sided [45.2 to 59.4], Standard Error of Mean 2.750
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% individually) with at least 99% statistical power, that 18 subjects were required to test for superiority for CLUE vision scores for Myopes; Test type: Superiority — A superiority Margin of 41 CLUE Points was used for Myopes; Mean Population Estimate = 63.3, 99% CI 2-sided [58.0 to 68.6], Standard Error of Mean 2.054

3. Primary Outcome: Proportion of Eyes With Unacceptable Lens Fitting
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope post lens insertion, the 1-week follow-up and any unscheduled visits. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The proportion of eyes with unacceptable lens fit was reported.
Time Frame: Up to 1-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 139
Number analyzed (Eyes) | 278
Proportion of eyes | 0
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.02 and an intraclass correlation of 0.70 with 2000 replicating trials, that 100 subjects were required to test for superiority to achieve a minimum statistical power of 90% with 95% central posterior credible; Test type: Superiority — A superiority margin of 0.05 was used; Bayesian beta- binomial model; Bayesian beta-binomial model for correlated binary data; Mean Proportion = 0.0019, 95% CI 2-sided [0.0000 to 0.0076], Standard Deviation 0.00209

4. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 1-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher was reported.
Time Frame: Up to 1-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Porportion of eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 139
Number analyzed (Eyes) | 278
Porportion of eyes | 0
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); [analysis description as in outcome 3, analysis 1]; Test type: Superiority — A superiority margin of 0.05 was used; Bayesian beta-binomial model; Bayesian beta-binomial model for correlated binary data; Mean Proportion = 0.0018, 95% CI 2-sided [0.0000 to 0.0078], Standard Deviation 0.00210

5. Secondary Outcome: CLUE Vision Score
Description: as for outcome 2
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 136
Units on a scale
  Hyperopes: number analyzed (Participants) | 49
  Hyperopes | 52.30 (19.121)
  Myopes: number analyzed (Participants) | 87
  Myopes | 63.27 (19.031)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% individually) with at least 80% statistical power, that 16 subjects were required to test for superiority for CLUE vision scores for Hyperopes; Test type: Superiority — A superiority Margin of 41 CLUE Points was used for Hyperopes; Mean Population Estimate = 52.3, 99% CI 2-sided [45.2 to 59.4], Standard Error of Mean 2.750
Statistical Analysis 2: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% individually) with at least 80% statistical power, that 15 subjects were required to test for superiority for CLUE vision scores for Myopes; Test type: Superiority — A superiority Margin of 46 CLUE Points was used for Myopes; Mean Population Estimate = 63.3, 99% CI 2-sided [58.0 to 68.6], Standard Error of Mean 2.054

6. Secondary Outcome: CLUE Comfort Score
Description: Subjective comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE comfort score was reported. The pre-specified aim was not to compare comfort between the hyperope and myope subgroups, therefore, comfort scores were reported for both groups combined.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 136
Units on a scale | 72.60 (20.696)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% individually) with at least 80% statistical power, that 11 subjects were required to test for superiority for CLUE comfort scores; Test type: Superiority — A Superiority margin of 52 CLUE points was used; Mean Population Estimate = 72.6, 99% CI 2-sided [68.1 to 77.1], Standard Error of Mean 1.763

7. Secondary Outcome: CLUE Handling Score
Description: Subjective Handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE handling score was reported. The pre-specified aim was not to compare comfort between the hyperope and myope subgroups, therefore, comfort scores were reported for both groups combined.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol with data collected at the 1-week follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 136
Units on a scale | 67.56 (20.619)
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a 2-sided one sample mean t-test with a family wise type I error rate of 5% (1% individually) with at least 80% statistical power, that 17 subjects were required to test for superiority for CLUE handling scores; Test type: Superiority — A Superiority margin of 53 CLUE points was used; Mean Population Estimate = 67.6, 99% CI 2-sided [63.0 to 72.1], Standard Error of Mean 1.770

8. Secondary Outcome: Proportion of Subject Achieving Optimal Lens Pair in 4 Lenses or Less
Description: The number of lenses to achieve the optimal pair for each subject was calculated as the original pair (2) plus all the required modifications to reach the optimal pair. In this study the minimum number of lenses per subject used was 2 where the maximum possible number of lenses used was 10. The data was dichotomized as Y=1 if the subject was able to achieve optimal lens pair in 4 lenses or lenses or less and 0 otherwise. A lens modification was performed if the subject reports unsatisfactory vision or was unable to obtain 20/30 distance visual acuity in both eyes. If the subject reported satisfactory vision with the lenses a modification was not required. However, based upon the investigator's findings on the measured visual acuity and/or over- refraction a modification may have been performed.
Time Frame: Up to 1-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of subjects
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 139
Proportion of subjects | 1
Statistical Analysis 1: Comparison: Test (Senofilcon A C3); It was calculated using a Bayesian beta-binomial model for correlated data with a reference rate of 0.98 and an intraclass correlation of 0.70 with 2000 replicating trials, that 92 subjects were required to test for superiority to achieve a minimum statistical power of 80% with 99% central posterior credible; Test type: Superiority — A superiority margin of 0.90 was used; Bayesian beta-binomial model; Bayesian beta-binomial model for correlated binary data; Mean Posterior Proportion = 0.985, 99% CI 2-sided [0.959 to 0.997], Standard Deviation 0.0071

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 7±3 days.
Groups:
- Test (Senofilcon A C3): Subjects that wore the Test (senofilcon A C3) lens during the study.
Arm/Group | Test (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/139
Serious Adverse Events (participants affected / at risk) | 0/139
Other Adverse Events (participants affected / at risk) | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT05222880/Prot_SAP_000.pdf